CLINICAL TRIAL: NCT01271712
Title: A Randomized, Double-blind, Placebo-controlled Phase III Study of Regorafenib Plus Best Supportive Care Versus Placebo Plus Best Supportive Care for Subjects With Metastatic and/or Unresectable Gastrointestinal Stromal Tumors (GIST) Whose Disease Has Progressed Despite Prior Treatment With at Least Imatinib and Sunitinib
Brief Title: Study of Regorafenib as a 3rd-line or Beyond Treatment for Gastrointestinal Stromal Tumors (GIST)
Acronym: GRID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14874; 2009-017957-37 (EudraCT Number)
Record Dates: First submitted 2010-12-17; First posted 2011-01-07 (Estimated); Results first posted 2013-10-25 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Gastrointestinal stromal cancer; GIST; multikinase inhibitor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — regorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Regorafenib (Stivarga, BAY73-4506) (Experimental): Participants received Regorafenib (Stivarga) 160 mg (4 x 40 mg tablets) per os once daily, 3 weeks on therapy followed by 1 week off therapy to comprise a cycle of 4 weeks
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506); Drug: Best supportive care
- Placebo (Placebo Comparator): Participants received matching Placebo tablets per os once daily, 3 weeks on therapy followed by 1 week off therapy to comprise a cycle of 4 weeks
  Interventions: Drug: Placebo; Drug: Best supportive care

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506) — 160 mg po once daily (od), 3 weeks on/1 week off. Route of administration: oral
  Arms: Regorafenib (Stivarga, BAY73-4506)
Drug: Placebo — once daily (od), 3 weeks on/1 week off. Route of administration: oral
  Arms: Placebo
Drug: Best supportive care — Best supportive care includes any method to preserve the comfort and dignity of the patients, and excludes any disease-specific anti-neoplastic therapy such as any kinase inhibitor, chemotherapy, radiation therapy, or surgical intervention.

SUMMARY:
A randomized, double-blind, placebo-controlled phase III study of regorafenib plus best supportive care versus placebo plus best supportive care for subjects with metastatic and/or unresectable gastrointestinal stromal tumors (GIST) whose disease has progressed despite prior treatment with at least imatinib and sunitinib.

The study is composed of 3 periods: A Screening Period, a Treatment Period, and a Survival Follow up Period.

Subjects randomized to be treated with regorafenib will receive 160 mg po od for 3 weeks of every 4 week (28 day) cycle (ie, 3 weeks on/1 week off). In addition subjects will receive best supportive care which excludes any disease specific anti cancer therapy such as any kinase inhibitor, chemotherapy, radiation therapy, or surgery.

Tumor assessment will be every 4 weeks for the first 3 months, every 6 weeks for the next 3 months (through month 6), and every 8 weeks until the end of treatment, or more frequently if clinically indicated. Tumor assessments include CT or MRI and will be performed until tumor progression is seen in a central radiology review.

Subjects receiving placebo who experience disease progression may be offered active treatment.

Subjects who experience progression during regorafenib treatment may continue open label treatment.

All subjects will enter the Survival Follow-up Period upon discontinuation of randomized study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 years of age.
* Subjects with histologically confirmed metastatic and/or unresectable GIST.
* At least imatinib and sunitinib as prior treatment regimens, with objective disease progression or intolerance to imatinib, as well as disease progression while on sunitinib therapy. Additionally, disease progression or intolerance to other systemic therapies, as well as investigational new agents, is allowed, except prior treatment with any other vascular endothelial growth factor receptor (VEGFR) inhibitor.
* Subjects must have at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1. A lesion in a previously irradiated area is eligible to be considered as measurable disease as long as there is objective evidence of progression of the lesion prior to study enrollment.

Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.

* Adequate bone marrow, liver, and renal function as assessed by laboratory parameters.

Recovery to NCI-CTCAE v4.0 Grade 0 or 1 level or recovery to baseline preceding the prior treatment from any previous drug/procedure-related toxicity (except alopecia and anemia).

Exclusion Criteria:

* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of study medication.
* Congestive heart failure New York Heart Association (NYHA) class 2.
* Unstable angina (angina symptoms at rest, new-onset angina, ie, within the last 3 months) or myocardial infarction (MI) within the past 6 months before start of study medication.
* Uncontrolled hypertension (systolic blood pressure 140 mmHg or diastolic pressure 90 mmHg despite optimal medical management).

Arterial thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), or pulmonary embolism within the 6 months before start of study drug or venous thrombotic events such as deep vein thrombosis within the 3 months before start of study drug.

* Ongoing infection grade 2 National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0.

Symptomatic metastatic brain or meningeal tumors.

* Subjects with evidence or history of bleeding diathesis. Any hemorrhage or bleeding event NCI-CTCAE version 4.0 grade 3 or higher within 4 weeks prior to the start of study drug.

Non-healing wound, ulcer, or bone fracture.

* Persistent proteinuria of NCI-CTCAE version 4.0 grade 3 or higher (3.5 g/24 hrs, measured by urine protein:creatinine ratio on a random urine sample).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2011-01-04 (Actual); Primary Completion 2012-01-26 (Actual); Study Completion 2019-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (55):
- United States (9):
  - Scottsdale, Arizona
  - Evanston, Illinois
  - Skokie, Illinois
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - New York, New York
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Seattle, Washington
- Austria (3):
  - Graz, Styria
  - Innsbruck
  - Vienna
- Leuven, Belgium
- Canada (3):
  - Edmonton, Alberta
  - London, Ontario
  - Toronto, Ontario
- China (4):
  - Guangzhou, Guangdong
  - Nanjing, Jiangsu
  - Beijing
  - Shanghai
- Helsinki, Finland
- France (4):
  - Bordeaux
  - Lille
  - Lyon
  - Villejuif
- Germany (7):
  - Mannheim, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - Bad Saarow, Brandenburg
  - Hanover, Lower Saxony
  - Cologne, North Rhine-Westphalia
  - Düsseldorf, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
- Tel Aviv, Israel
- Italy (4):
  - Bologna, Emilia-Romagna
  - Milan, Lombardy
  - Turin, Piedmont
  - Palermo, Sicily
- Japan (6):
  - Nagoya, Aichi-ken
  - Kashiwa, Chiba
  - Sapporo, Hokkaido
  - Chuo-ku, Tokyo
  - Niigata
  - Osaka
- Netherlands (2):
  - Leiden
  - Nijmegen
- Warsaw, Poland
- Singapore, Singapore
- South Korea (3):
  - Goyang-si, Gyeonggido
  - Busan
  - Seoul
- Spain (2):
  - L'Hospitalet de Llobregat, Barcelona
  - Barcelona
- United Kingdom (3):
  - Leicester, Leicestershire
  - London
  - Manchester

REFERENCES:
- [Result] Demetri GD, Reichardt P, Kang YK, Blay JY, Rutkowski P, Gelderblom H, Hohenberger P, Leahy M, von Mehren M, Joensuu H, Badalamenti G, Blackstein M, Le Cesne A, Schoffski P, Maki RG, Bauer S, Nguyen BB, Xu J, Nishida T, Chung J, Kappeler C, Kuss I, Laurent D, Casali PG; GRID study investigators. Efficacy and safety of regorafenib for advanced gastrointestinal stromal tumours after failure of imatinib and sunitinib (GRID): an international, multicentre, randomised, placebo-controlled, phase 3 trial. Lancet. 2013 Jan 26;381(9863):295-302. doi: 10.1016/S0140-6736(12)61857-1. Epub 2012 Nov 22. PMID 23177515
- [Result] Poole CD, Connolly MP, Chang J, Currie CJ. Health utility of patients with advanced gastrointestinal stromal tumors (GIST) after failure of imatinib and sunitinib: findings from GRID, a randomized, double-blind, placebo-controlled phase III study of regorafenib versus placebo. Gastric Cancer. 2015 Jul;18(3):627-34. doi: 10.1007/s10120-014-0391-x. Epub 2014 Jun 24. PMID 24957256
- [Result] Komatsu Y, Doi T, Sawaki A, Kanda T, Yamada Y, Kuss I, Demetri GD, Nishida T. Regorafenib for advanced gastrointestinal stromal tumors following imatinib and sunitinib treatment: a subgroup analysis evaluating Japanese patients in the phase III GRID trial. Int J Clin Oncol. 2015 Oct;20(5):905-12. doi: 10.1007/s10147-015-0790-y. Epub 2015 Feb 6. PMID 25655899
- [Derived] Mross K, Frost A, Steinbild S, Hedbom S, Buchert M, Fasol U, Unger C, Kratzschmar J, Heinig R, Boix O, Christensen O. A phase I dose-escalation study of regorafenib (BAY 73-4506), an inhibitor of oncogenic, angiogenic, and stromal kinases, in patients with advanced solid tumors. Clin Cancer Res. 2012 May 1;18(9):2658-67. doi: 10.1158/1078-0432.CCR-11-1900. Epub 2012 Mar 15. PMID 22421192
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 240 participants with metastatic and/or unresectable GIST whose disease had progressed despite prior treatments with at least imatinib and sunitinib were screened; 199 were randomized. Patients must have shown objective disease progression or intolerance to imatinib, as well as disease progression while on sunitinib treatment.
Pre-assignment Details: Participants were randomized in a 2:1 ratio to receive either regorafenib (133 patients) or placebo (66 patients). Randomization was stratified according 3rd vs. 4th line of therapy (at least 50% of patients were to be 3rd line), and geographical region (Asia vs.rest of world).
Groups:
- Placebo First, Then Option of Open Label Regorafenib Treatment: Double blind phase: participants received matching Placebo tablets per os once daily, 3 weeks on therapy followed by 1 week off therapy to comprise a cycle of 4 weeks. Open Label phase: participants on placebo who switched to Regorafenib, received Regorafenib 160 mg (4 x 40 mg tablets) per os once daily, 3 weeks on therapy followed by 1 week off therapy to comprise a cycle of 4 weeks.
Period: Double Blind Treatment
Arm/Group | Regorafenib (Stivarga, BAY73-4506) | Placebo First, Then Option of Open Label Regorafenib Treatment
Started | 133 | 66
Participants Received Treatment | 132 | 66
Completed | 91 (91 participants started open-label treatment with regorafenib) | 58 (58 participants started open-label treatment with regorafenib)
Not Completed | 42 | 8
Not completed — Death | 2 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Adverse Event | 9 | 4
Not completed — Progressive disease | 23 | 3
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Non compliance with study drug | 2 | 0
Not completed — receive no study drug | 1 | 0
Period: Open Label Treatment
Arm/Group | Regorafenib (Stivarga, BAY73-4506) | Placebo First, Then Option of Open Label Regorafenib Treatment
Started | 91 | 58
Completed | 0 | 0
Not Completed | 91 | 58
Not completed — Death | 6 | 5
Not completed — Withdrawal by Subject | 6 | 11
Not completed — Physician Decision | 2 | 0
Not completed — Adverse Event | 14 | 8
Not completed — Progressive disease | 59 | 32
Not completed — transferred to rollover study | 1 | 0
Not completed — Non-compliance with study drug | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Switching to other therapy | 2 | 1
Period: Safety Follow-up
Arm/Group | Regorafenib (Stivarga, BAY73-4506) | Placebo First, Then Option of Open Label Regorafenib Treatment
Started | 118 (All participants who discontinued study drug entered 30-day Safety Follow-up) | 52 (All participants who discontinued study drug entered 30-day Safety Follow-up)
Completed | 97 | 37
Not Completed | 21 | 15
Not completed — Death | 11 | 7
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Not analyzed after cutoff 08Jun2015 | 3 | 4
Not completed — No follow-up | 1 | 1
Not completed — Progressive disease | 1 | 0
Period: Survival Follow-up
Arm/Group | Regorafenib (Stivarga, BAY73-4506) | Placebo First, Then Option of Open Label Regorafenib Treatment
Started | 100 (All participants entered Survival Follow-up immediately after safety follow-up) | 39 (All participants entered Survival Follow-up immediately after safety follow-up)
Completed | 85 (85 participants died and completed survival follow-up.) | 33 (33 participants died and completed survival follow-up.)
Not Completed | 15 | 6
Not completed — Not analyzed after cutoff 08Jun2015 | 15 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regorafenib (Stivarga, BAY73-4506) | Placebo | Total
Number analyzed (Participants) | 133 | 66 | 199
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.2 (12.5) | 58.1 (13.9) | 58.2 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 24 | 72
  Male | 85 | 42 | 127
ECOG Performance Status (PS)] [Count of Participants; unit: Participants] — ECOG = Eastern cooperative oncology group PS levels are 0 (Fully active, able to carry on all pre-disease performance), 1 (ambulatory and able to carry out work of a light or sedentary), 2 (Ambulatory and capable of all selfcare but unable to carry out any work activities), 3 (Capable of only limited selfcare, confined to bed or chair more than 50% of awake time), 4 (Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair) and 5 (death).
  Participants
    PS 0 | 73 | 37 | 110
    PS 1 | 60 | 29 | 89
    PS 2 | 0 | 0 | 0
    Missing | 0 | 0 | 0
Prior anti-cancer drug group [Count of Participants; unit: Participants] — 3rd line: 3rd in sequence of multiple therapies: imatinib (1st); sunitinib (2nd). 4th line and beyond: 4th in sequence of multiple therapies: imatinib (1st); sunitinib (2nd); other (3rd).
  Participants
    3rd line | 74 | 39 | 113
    4th line and beyond | 59 | 27 | 86

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free Survival (PFS) was defined as the time from date of randomization to radiological disease progression or death due to any cause, whichever occurs first. PFS was based on central radiological assessment using modified RECIST (Response Evaluation Criteria in Solid Tumors) v.1.1. Progression is defined as at least a 20% increase in the sum of diameters of target lesions taking as reference the smallest sum on study; or unequivocal progression of existing non-target lesions; or appearance of new lesions. Subjects without progression or death at the time of analysis were censored at their last date of tumor evaluation. Results are based on central evaluation.
Time Frame: From randomization of the first subject until approximately 144 progression-free survival events had occurred (study duration approximately one year)
Population: Full Analysis Set (FAS) - defined as all randomized participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Regorafenib (Stivarga, BAY73-4506) | Placebo
Number analyzed (Participants) | 133 | 66
Days | 147 [122 to 173] | 28 [28 to 32]
Statistical Analysis 1: Comparison: Regorafenib (Stivarga, BAY73-4506) vs Placebo; The two treatment groups were compared using a stratified log rank test with a one-sided alpha of 0.01 stratified by (3rd vs 4th-line; and geographical region). The null hypothesis that both treatment arms have the same PFS distribution was tested against the alternative hypothesis that the distribution of PFS in the regorafenib arm is different from the control arm according to a proportional hazards relation between the treatment arms; Test type: Superiority or Other; p < 0.000001, Log Rank; stratified
Statistical Analysis 2: Comparison: Regorafenib (Stivarga, BAY73-4506) vs Placebo; Hazard ratio and its 95% CI (Confidence Interval) was based on stratified Cox Regression Model; Test type: Superiority or Other; Regression, Cox; stratified; Hazard Ratio (HR) = 0.268, 95% CI 2-sided [0.185 to 0.388] — regorafenib over placebo

2. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) was defined as the time from date of randomization to death due to any cause. Subjects still alive at the time of analysis were censored at their date of last contact. Median OS was not observed at the time of PFS analysis and first analysis of OS, therefore only the proportion of death events was reported in the results posting system. This approach was maintained for the subsequent updates in the results posting system.
Time Frame: From randomization of the first subject until date of database cutoff (08 Jun 2015)
Population: Full Analysis Set (FAS). 58 (87.9%) patients in placebo group and 91 (68.4%) patients in regorafenib had started open-label treatment with regorafenib before time of final database cutoff 08 Jun 2015
Measure: Number; unit: Percentage of patients with death
Arm/Group | Regorafenib (Stivarga, BAY73-4506) | Placebo
Number analyzed (Participants) | 133 | 66
Percentage of patients with death | 82.0 | 80.3
Statistical Analysis 1: Comparison: Regorafenib (Stivarga, BAY73-4506) vs Placebo; Test type: Superiority or Other; p = 0.285777, Log Rank; stratified
Statistical Analysis 2: Comparison: Regorafenib (Stivarga, BAY73-4506) vs Placebo; Hazard ratio and its 95% CI was based on stratified Cox Regression Model; Test type: Superiority or Other; Regression, Cox; stratified; Hazard Ratio (HR) = 0.909, 95% CI 2-sided [0.653 to 1.265] — regorafenib over control. 58 (87.9%) patients in placebo group and 91 (68.4%) patients in regorafenib had started open-label treatment with regorafenib before time of final database cutoff 08 Jun 2015

3. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression (TTP) was defined as the time from date of randomization to disease progression (based on central radiological assessment using modified RECIST [Response Evaluation Criteria in Solid Tumors] v.1.1). Progression is defined as at least a 20% increase in the sum of diameters of target lesions taking as reference the smallest sum on study; or unequivocal progression of existing non-target lesions; or appearance of new lesions. Subjects without progression at the time of analysis were censored at their last date of tumor evaluation. Results are based on central evaluation.
Time Frame: From randomization of the first subject until until date of database cutoff (26 Jan 2012); study duration approximately 1 year
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Regorafenib (Stivarga, BAY73-4506) | Placebo
Number analyzed (Participants) | 133 | 66
Days | 165 [125 to 174] | 28 [28 to 34]
Statistical Analysis 1: Comparison: Regorafenib (Stivarga, BAY73-4506) vs Placebo; Test type: Superiority or Other; p < 0.000001, Log Rank; stratified
Statistical Analysis 2: Comparison: Regorafenib (Stivarga, BAY73-4506) vs Placebo; Test type: Superiority or Other; Regression, Cox; stratified; Hazard Ratio (HR) = 0.248, 95% CI 2-sided [0.170 to 0.364]

4. Secondary Outcome: Tumor Response
Description: Tumor Response of a subject was defined as the best tumor response (Complete Response [CR: disappearance of all clinical and radiological evidence of tumor (both target and non-target).], Partial Response [PR: at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum, no unequivocal progression of existing non-target lesions, and no appearance of new lesions.], Stable Disease [SD: steady state of disease. Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, no unequivocal progression of existing non-target lesions, and no appearance of new lesions.], or Progressive Disease [PD: at least a 20% increase in the sum of diameters of target lesions taking as reference the smallest sum on study or unequivocal progression of existing non-target lesions, or appearance of new lesions.]) observed during the trial period and assessed according to RECIST v1.1 criteria. Results are based on central evaluation.
Time Frame: From randomization of the first subject until date of database cutoff (26 Jan 2012); study duration approximately 1 year
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Regorafenib (Stivarga, BAY73-4506) | Placebo
Number analyzed (Participants) | 133 | 66
Percentage of Participants
  Complete Response (CR) | 0 [0 to 0] | 0 [0 to 0]
  Partial Response (PR) | 4.5 [1.7 to 9.6] | 1.5 [0 to 8.2]
  Stable Disease (SD) | 71.4 [63.0 to 78.9] | 33.3 [22.2 to 46.0]
  Progressive Disease (PD) | 21.1 [14.5 to 29.0] | 63.6 [50.9 to 75.1]
  Not Assessable | 3.0 [0.8 to 7.5] | 1.5 [0 to 8.2]

5. Secondary Outcome: Objective Response Rate
Description: Objective response rate was defined as the percentage of subjects whose best response was Complete Response (CR: disappearance of all clinical and radiological evidence of tumor (both target and non-target).) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum, no unequivocal progression of existing non-target lesions, and no appearance of new lesions.) according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1). Results are based on central evaluation.
Time Frame: as for outcome 4
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Regorafenib (Stivarga, BAY73-4506) | Placebo
Number analyzed (Participants) | 133 | 66
Percentage of Participants | 4.5 [1.7 to 9.6] | 1.5 [0.0 to 8.2]

6. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease Control Rate (DCR) was defined as the percentage of subjects whose best response was Complete Response (CR: disappearance of all clinical and radiological evidence of tumor (both target and non-target).), Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum, no unequivocal progression of existing non-target lesions, and no appearance of new lesions.), or Stable Disease (SD: steady state of disease. Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, no unequivocal progression of existing non-target lesions, and no appearance of new lesions.) according to RECIST v1.1 criteria. SD had to be maintained for at least 12 weeks from the first demonstration of that rating. Results are based on central evaluation.
Time Frame: as for outcome 4
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Regorafenib (Stivarga, BAY73-4506) | Placebo
Number analyzed (Participants) | 133 | 66
Percentage of Participants | 52.6 [43.8 to 61.3] | 9.1 [3.4 to 18.7]

7. Secondary Outcome: Duration of Response (DOR)
Description: Duration of Response was defined as the time from date of first response (Complete Response [CR: disappearance of all clinical and radiological evidence of tumor (both target and non-target).] or Partial Response [PR: at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum, no unequivocal progression of existing non-target lesions, and no appearance of new lesions.]) to the date when Progressive Disease (PD: at least a 20% increase in the sum of diameters of target lesions taking as reference the smallest sum on study or unequivocal progression of existing non-target lesions, or appearance of new lesions.) is first documented, or to the date of death, whichever occurs first, according to RECIST v1.1. Subjects still having CR or PR and have not died at the time of analysis were censored at their last date of tumor evaluation. Duration of response defined for responders only, i.e CR or PR. Results are based on central evaluation.
Time Frame: as for outcome 4
Population: Full Analysis Set with response participants
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Regorafenib (Stivarga, BAY73-4506) | Placebo
Number analyzed (Participants) | 6 | 1
Days | 99 [42 to NA] — A complete confidence interval (CI) cannot be calculated because there are too few patients in the data set. | 30 [NA to NA] — CI cannot be calculated because there is only 1 patient in the data set.

ADVERSE EVENTS:
Time Frame: From first administration of treatment till 30 days after last dose of treatment.
Description: At primary completion (cutoff 26JAN2012) blinded patients who received either regorafenib or placebo were reported in "Regorafenib (DoubleBlindOnly)" and "Placebo (DoubleBlindOnly)" respectively; patients who received regorafenib after unblinding were reported in "Placebo, OpenLabelOnly(Switch to Regorafenib)". This safety update (cutoff 15APR2019) was reported in "Treated with Regorafenib at any time" and "Treated with Regorafenib for>1 year".
Groups:
- Regorafenib (Double Blind Only): Participants received Regorafenib (Stivarga) 160 mg (4 x 40 mg tablets) per os once daily, 3 weeks on therapy followed by 1 week off therapy to comprise a cycle of 4 weeks
- Placebo (Double Blind Only): Participants received matching Placebo tablets per os once daily, 3 weeks on therapy followed by 1 week off therapy to comprise a cycle of 4 weeks
- Placebo, Open Label Only (Switch to Regorafenib): Participants switched to Open-label Regorafenib treatment from Placebo. Participants received Regorafenib (Stivarga) 160 mg (4 x 40 mg tablets) per os once daily, 3 weeks
- Treated With Regorafenib at Any Time: Treated with Regorafenib at any time: At any time, participants received Regorafenib (Stivarga) 160 mg (4 x 40 mg tablets) per os once daily, 3 weeks on therapy followed by 1 week off therapy to comprise a cycle of 4 weeks
- Treated With Regorafenib for > 1 Year: Treated with Regorafenib for > 1 year: For more than a year, participants received Regorafenib (Stivarga) 160 mg (4 x 40 mg tablets) per os once daily, 3 weeks on therapy followed by 1 week off therapy to comprise a cycle of 4 weeks
Arm/Group | Regorafenib (Double Blind Only) | Placebo (Double Blind Only) | Placebo, Open Label Only (Switch to Regorafenib) | Treated With Regorafenib at Any Time | Treated With Regorafenib for > 1 Year
All-Cause Mortality (participants affected / at risk) | 40/41 | 7/8 | 47/58 | 155/190 | 48/75
Serious Adverse Events (participants affected / at risk) | 23/41 | 8/8 | 31/58 | 103/190 | 39/75
Other Adverse Events (participants affected / at risk) | 40/41 | 7/8 | 58/58 | 189/190 | 75/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib (Double Blind Only) (N=41) | Placebo (Double Blind Only) (N=8) | Placebo, Open Label Only (Switch to Regorafenib) (N=58) | Treated With Regorafenib at Any Time (N=190) | Treated With Regorafenib for > 1 Year (N=75)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 0 (0)
Congenital, familial and genetic disorders - Other (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 6 (6)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Conduction disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac disorders - Other (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 0 (0) | 2 (2) | 9 (10) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (4) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 2 (3)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritoneal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Death NOS (General disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 2 (2)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Fatigue (General disorders) | 2 (4) | 1 (2) | 2 (2) | 5 (7) | 2 (2)
Fever (General disorders) | 1 (1) | 0 (0) | 2 (2) | 5 (5) | 2 (2)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other (General disorders) | 1 (1) | 1 (1) | 2 (3) | 5 (6) | 3 (3)
Pain (General disorders) | 1 (1) | 0 (0) | 2 (3) | 3 (4) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 1 (2) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Hepatic hemorrhage (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 3 (6) | 1 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Creatinine increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
INR increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Investigations - Other (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (2)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 1 (2)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 8 (9) | 3 (4)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 4 (5) | 3 (4)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoglossal nerve disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 3 (3) | 6 (6) | 3 (3)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (4) | 3 (5) | 1 (1)
Eye disorders - Other (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Mania (Psychiatric disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Psychiatric disorders - Other (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (2) | 4 (5) | 1 (1)
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (2)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Surgical and medical procedures - Other (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 2 (2)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular disorders - Other (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral ischemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 1 (2) | 4 (5) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib (Double Blind Only) (N=41) | Placebo (Double Blind Only) (N=8) | Placebo, Open Label Only (Switch to Regorafenib) (N=58) | Treated With Regorafenib at Any Time (N=190) | Treated With Regorafenib for > 1 Year (N=75)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 7 (7) | 5 (5)
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 4 (4) | 7 (7) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 4 (7) | 0 (0) | 11 (25) | 35 (77) | 17 (35)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (9) | 6 (17) | 4 (9)
Hypothyroidism (Endocrine disorders) | 4 (4) | 0 (0) | 6 (6) | 39 (50) | 25 (32)
Abdominal pain (Gastrointestinal disorders) | 14 (18) | 0 (0) | 16 (23) | 62 (122) | 26 (60)
Ascites (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 6 (8) | 1 (3)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 7 (10) | 6 (9)
Constipation (Gastrointestinal disorders) | 10 (14) | 5 (6) | 16 (30) | 63 (101) | 28 (52)
Diarrhea (Gastrointestinal disorders) | 15 (20) | 1 (1) | 24 (67) | 96 (353) | 53 (281)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 1 (2) | 6 (9) | 19 (39) | 11 (30)
Dry mouth (Gastrointestinal disorders) | 5 (5) | 0 (0) | 5 (6) | 15 (16) | 5 (6)
Flatulence (Gastrointestinal disorders) | 4 (4) | 0 (0) | 3 (3) | 10 (11) | 5 (6)
Mucositis oral (Gastrointestinal disorders) | 14 (18) | 2 (3) | 21 (48) | 81 (174) | 38 (111)
Nausea (Gastrointestinal disorders) | 9 (12) | 3 (4) | 18 (33) | 61 (110) | 32 (66)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 4 (4) | 0 (0) | 4 (7) | 17 (21) | 11 (15)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 7 (7) | 5 (5)
Vomiting (Gastrointestinal disorders) | 10 (11) | 3 (5) | 12 (24) | 48 (85) | 21 (54)
Chills (General disorders) | 1 (1) | 0 (0) | 4 (4) | 11 (19) | 8 (16)
Edema limbs (General disorders) | 3 (4) | 3 (3) | 11 (20) | 33 (72) | 17 (53)
Fatigue (General disorders) | 18 (32) | 3 (4) | 32 (83) | 104 (251) | 46 (137)
Fever (General disorders) | 10 (17) | 1 (1) | 18 (24) | 52 (83) | 25 (46)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 3 (3) | 18 (22) | 14 (17)
Localized edema (General disorders) | 2 (2) | 1 (1) | 3 (5) | 8 (10) | 5 (7)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 7 (8) | 6 (7)
General disorders and administration site conditions - Other (General disorders) | 1 (1) | 0 (0) | 4 (5) | 10 (11) | 5 (6)
Pain (General disorders) | 5 (8) | 1 (1) | 19 (46) | 55 (115) | 29 (73)
Alanine aminotransferase increased (Investigations) | 4 (9) | 1 (2) | 6 (15) | 20 (41) | 4 (10)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 3 (6) | 11 (21) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 4 (9) | 2 (2) | 8 (15) | 23 (58) | 6 (24)
Blood bilirubin increased (Investigations) | 4 (6) | 1 (3) | 9 (15) | 22 (52) | 7 (27)
GGT increased (Investigations) | 0 (0) | 1 (2) | 2 (2) | 4 (4) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 3 (11) | 6 (19) | 3 (14)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 6 (8) | 13 (25) | 6 (12)
Investigations - Other (Investigations) | 0 (0) | 0 (0) | 2 (14) | 14 (49) | 10 (28)
Platelet count decreased (Investigations) | 1 (5) | 0 (0) | 6 (25) | 15 (46) | 10 (34)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 6 (17) | 4 (15)
Weight gain (Investigations) | 0 (0) | 1 (1) | 2 (3) | 3 (4) | 2 (3)
Weight loss (Investigations) | 4 (5) | 2 (2) | 11 (20) | 40 (72) | 22 (44)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 4 (4)
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 11 (12) | 9 (10)
Infections and infestations - Other (Infections and infestations) | 2 (3) | 0 (0) | 5 (7) | 21 (39) | 13 (26)
Rash pustular (Infections and infestations) | 2 (2) | 0 (0) | 2 (17) | 13 (49) | 10 (42)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 6 (6) | 5 (5)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (4) | 6 (7) | 4 (4)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 5 (5)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 9 (12) | 26 (41) | 21 (36)
Urinary tract infection (Infections and infestations) | 2 (3) | 0 (0) | 2 (4) | 12 (17) | 6 (9)
Anorexia (Metabolism and nutrition disorders) | 15 (21) | 3 (5) | 20 (42) | 77 (134) | 32 (72)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 5 (5) | 6 (8) | 4 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 3 (3) | 9 (10) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 3 (8) | 9 (15) | 4 (4)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 12 (18) | 20 (31) | 13 (22)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 3 (4) | 8 (11) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 10 (13) | 5 (7)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3) | 4 (4) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 5 (5) | 13 (18) | 9 (10)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 7 (7) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 4 (7) | 14 (20) | 8 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 4 (6) | 21 (29) | 14 (20)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 5 (9) | 5 (9)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 4 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 4 (7) | 6 (14) | 3 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 10 (17) | 34 (76) | 17 (49)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 4 (5) | 14 (17) | 10 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (2) | 7 (15) | 28 (51) | 17 (37)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 6 (16) | 6 (16)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0) | 4 (4) | 17 (19) | 9 (11)
Headache (Nervous system disorders) | 4 (4) | 0 (0) | 11 (21) | 37 (72) | 23 (55)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 3 (5) | 11 (19) | 9 (13)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (7) | 0 (0) | 4 (8) | 16 (22) | 6 (7)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1) | 3 (4) | 7 (9) | 2 (2)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 7 (7) | 7 (7)
Eye disorders - Other (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (6) | 4 (4)
Anxiety (Psychiatric disorders) | 4 (4) | 0 (0) | 3 (4) | 9 (10) | 4 (5)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2) | 10 (11) | 4 (5)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1) | 3 (4) | 21 (22) | 14 (15)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 11 (18) | 27 (44) | 15 (32)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 0 (0) | 7 (9) | 22 (32) | 11 (16)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (6) | 10 (15) | 7 (10)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 0 (0) | 9 (11) | 42 (71) | 17 (36)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 5 (5) | 4 (4)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 11 (12) | 28 (32) | 14 (17)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (3) | 7 (9) | 3 (3)
Renal and urinary disorders - Other (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 10 (12) | 4 (5)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 6 (11) | 23 (58) | 9 (21)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 7 (8) | 4 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (9) | 0 (0) | 21 (26) | 62 (84) | 33 (49)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 2 (3) | 13 (15) | 7 (8)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (3) | 10 (17) | 7 (12)
Erythroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (5) | 9 (11) | 6 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 2 (2) | 6 (11) | 4 (9)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 7 (10) | 27 (41) | 17 (28)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 9 (39) | 6 (36)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 17 (37) | 1 (1) | 39 (151) | 126 (666) | 58 (455)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (2) | 7 (8) | 20 (27) | 10 (15)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 3 (3) | 12 (12) | 7 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (7) | 0 (0) | 8 (10) | 32 (71) | 16 (26)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 7 (8) | 4 (5)
Hypertension (Vascular disorders) | 18 (32) | 3 (3) | 37 (97) | 124 (697) | 62 (552)
Thromboembolic event (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 6 (7) | 5 (5)

LIMITATIONS AND CAVEATS:
Overall survival results are confounded by the fact that 85% of the participants initially randomized to placebo switched to open-label regorafenib.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days